CLINICAL TRIAL: NCT06100952
Title: A Multicenter, Randomized, Double-Masked, Sham-Controlled, Parallel-Group Phase 3 Study to Evaluate the Efficacy and Safety of Epithelium-On Corneal Cross-linking in Subjects 8 to 45 Years of Age with Keratoconus (APRICITY-B)
Brief Title: Epithelium-On Corneal Cross-linking in Subjects 8 to 45 Years of Age with Keratoconus
Acronym: Apricity-B
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Epion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXL-006-B
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Treatment (Experimental): Epithelium-on corneal cross-linking
  Interventions: Combination Product: Riboflavin and Sodium Iodide solution and Ultraviolet-A treatment
- Control Treatment (Placebo Comparator): Placebo and sham for epithelium-on corneal cross-linking
  Interventions: Combination Product: Placebo and sham treatment

INTERVENTIONS:
Combination Product: Riboflavin and Sodium Iodide solution and Ultraviolet-A treatment — Drug: Ribostat riboflavin and sodium iodide ophthalmic solution
  Device: UV-3000 ultraviolet A light source
  Arms: Active Treatment
Combination Product: Placebo and sham treatment — Drug: placebo ophthalmic solution
  Device: UV-3000 light source
  Arms: Control Treatment

SUMMARY:
A Multicenter, Randomized, Double-Masked, Sham-Controlled, Parallel-Group Phase 3 Study to Evaluate the Efficacy and Safety of Epithelium-On Corneal Cross-linking in Subjects 8 to 45 Years of Age With Keratoconus

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus

Exclusion Criteria:

* Minimal corneal thickness < 350 microns
* Non-keratoconic ectatic disease
* Contraindications or hypersensitivities to any required study medications
* Pregnancy or breastfeeding
* Certain concomitant ocular conditions

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Best Spectacle-Corrected Distance Visual Acuity (BSCDVA) | Baseline to 12 months
  BSCDVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts. The score ranges from 0 to 100, with a higher score representing better visual functioning.

SECONDARY OUTCOMES:
Vision-related Quality of Life as Assessed by the National Eye Institute 25-Item Visual Function Questionnaire (NEI-VFQ-25) | Baseline to 12 months
  The score on the NEI-VFQ-25 ranges from 0 to 100, with a higher score indicating greater functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Belin, MD, Study Director — Epion Therapeutics
Locations (12):
- United States (12):
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Catalina Eye Center, Tucson, Arizona
  - Inland Eye Specialists, Murrieta, California
  - University of Colorado, Aurora, Colorado
  - Chicago Cornea Consultants, Highland Park, Illinois
  - Claris Vision LLC Eye Health Vision Centers - Dartmouth, North Dartmouth, Massachusetts
  - Truhlsen Eye Institute, Omaha, Nebraska
  - Providence Eye and Laser Specialists, Charlotte, North Carolina
  - VRF Eye Specialty Group, Memphis, Tennessee
  - Dell Laser Consultants, Austin, Texas
  - Hoopes Vision, Draper, Utah
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No